CLINICAL TRIAL: NCT02921386
Title: A Phase 2 Study of the Effect of Meals With Various Amounts of Fat Given Immediately After Dosing on the Pharmacokinetics of an Oral Testosterone Undecanoate
Brief Title: The Effect of Various Amounts of Fat on PK of Oral Testosterone Undecanoate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CLAR-16015
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Results first posted 2018-04-12 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, 5-period crossover food effect study
Oversight: Data Monitoring Committee: No

ARMS (5):
- Breakfast A - Fasting (Other): Oral Testosterone Undecanoate 237 mg administered twice daily immediately prior to Fasting at breakfast and immediately prior to dinner.
  Interventions: Drug: Oral Testosterone Undecanoate
- Breakfast B - 15 g fat (Other): Oral Testosterone Undecanoate 237 mg administered twice daily immediately prior to 15 g fat breakfast and immediately prior to dinner.
  Interventions: Drug: Oral Testosterone Undecanoate
- Breakfast C - 30 g fat (Other): Oral Testosterone Undecanoate 237 mg administered twice daily immediately prior to 30 g fat breakfast and immediately prior to dinner.
  Interventions: Drug: Oral Testosterone Undecanoate
- Breakfast D - 45 g fat (Other): Oral Testosterone Undecanoate 237 mg administered twice daily immediately prior to 45 g fat breakfast and immediately prior to dinner.
  Interventions: Drug: Oral Testosterone Undecanoate
- Breakfast E - High Fat (Other): Oral Testosterone Undecanoate 237 mg administered twice daily immediately prior to high fat breakfast and immediately prior to dinner.
  Interventions: Drug: Oral Testosterone Undecanoate

INTERVENTIONS:
Drug: Oral Testosterone Undecanoate — All study participants received Oral TU dose of 237 mg TU twice daily before breakfast and dinner for 14 days and throughout 5 crossover periods

SUMMARY:
A Phase 2, open-label, randomized, cross-over, pharmacokinetic study designed to determine the effect of meals of various amounts of fat given immediately prior to dosing on the pharmacokinetics of oral testosterone undecanoate. Approximately 20 hypogonadal subjects will be dosed for a 14 day run-in period. This will be followed by a randomized sequence of five periods over a 6 day confinement period. Subjects will receive a randomly ordered sequence of breakfast meals containing various amounts of fat, fasting, 15 g, 30 g, 45 g and a high fat breakfast consistent Guidance for Industry on Food-Effect Bioavailability and Fed Bioequivalence Studies.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, randomized, cross over, pharmacokinetic study. Subjects will initially be dosed for 2 weeks (Run-In Phase) to allow suppression of endogenous testosterone production, while allowing the oral TU to reach steady state. The subjects will then be confined to a clinical unit in which they undergo the PK Phase of the study. During the PK Phase of the study, subjects will undergo a five-period cross-over in which oral TU is dosed twice daily. Subjects will dose in the morning and in the evening immediately prior to protocol-defined meals. The protocol-defined breakfasts will contain various levels of fat including 15 g, 30 g, 45 g, a breakfast consistent with the fat and calorie content of the high-fat breakfast consistent with recommendations in the Guidance for Industry on Food-Effect Bioavailability and Fed Bioequivalence Studies (December 2002), or while fasting (with no meal until 4 hours post-dose). Subjects will be randomized to a designated sequence of the protocol-defined breakfasts, or the fasted state. The subjects will be required to consume the entire breakfast within 20 minutes during the PK Phase. The protocol-defined evening meal will be required to be consumed within 20 minutes. The 5 meal periods will occur on sequential days.

Approximately twenty (20) subjects will be enrolled in order to ensure completion of 16 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Man 18 to 65 years of age, inclusive, with a clinical diagnosis of hypogonadism (signs/symptoms consistent with hypogonadism for testosterone naïve subjects and history of signs/symptoms for subjects who have received prior treatment) as well as testosterone levels consistent with hypogonadism as defined by 2 morning total T values of <300 ng/dL (between 6:00 and 10:00 AM drawn on 2 separate days [approximately 7 (±2) days apart].
2. Adequate venous access in the left or right arm to allow collection of a number of blood samples via a venous cannula.
3. Must be naïve to androgen-replacement therapy or washed out of prior androgen replacement therapies; that is, be willing to cease current T treatment or currently not be taking T treatment, (washout durations specified in exclusion criterion #1). Subjects must remain off all forms of T, except for dispensed study drug, throughout the entire study.
4. Subjects on replacement therapy for hypopituitarism or multiple endocrine deficiencies must be on stable doses of thyroid hormone and adrenal replacement hormones for at least 14 days before Screen 1.
5. Has voluntarily given written informed consent to participate in this study.

Exclusion Criteria:

1. Received oral topical (eg, gel or patch), intranasal, or buccal T therapy within the previous 2 weeks, intramuscular T injection of short-acting duration (eg, T enanthate, T cypionate) within the previous 4 weeks, intramuscular T injection of long-acting duration (eg, AVEED) within the previous 20 weeks, or T implantable pellets (Testopel®) within the previous 6 months.
2. Has an intercurrent disease deemed clinically significant in the opinion of the investigator of any type; in particular, liver, kidney, uncontrolled or poorly controlled heart disease, including hypertension, congestive heart failure or coronary heart disease, or psychiatric-illness, including severe depression.
3. Has had a recent (within 2 years) history of stroke, transient ischemic attack, or acute coronary event.
4. Has a mean of the triplicate assessment of sBP > 150 mm Hg and/or dBP > 90 mm Hg at screening (if prescribed antihypertensives, subject should be taking medications on the day of the screening visit with a sip of water). Subjects < 60 years of age and prescribed antihypertensives will be excluded if the mean of the triplicate assessment of sBP > 140 mm Hg and/or dBP > 90 mm Hg at screening.
5. Has had recent (within 2 years) history of angina or stent (coronary or carotid) placement.
6. Has untreated, severe obstructive sleep apnea.
7. Has clinically significant abnormal laboratory values, including serum transaminases > 2 × upper limits of normal (ULN), serum bilirubin > 1.5 × ULN and serum creatinine > 1.5 × ULN.
8. Has a hematocrit (HCT) value of < 35% or > 48%.
9. Has a history of polycythemia, either idiopathic or associated with TRT treatment.
10. Is a diabetic subject with a glycosylated hemoglobin > 8.5%.
11. Has a body mass index (BMI) ≥ 38 kg/m2.
12. Has been on stable doses of antihypertensive medication for < 3 months.
13. Has an abnormal prostate digital rectal examination [(DRE); palpable nodules], elevated PSA (serum PSA > 4.0 ng/mL), I-PSS > 19 points at screening, and/or history of, or current or suspected, prostate cancer.
14. Has a history of, or current or suspected, breast cancer.
15. Has a history of abnormal bleeding tendencies or thrombophlebitis unrelated to venipuncture or intravenous cannulation within the previous 2 years.
16. Use of dietary supplements such as saw palmetto or phytoestrogens and any dietary supplements that may increase total T, such as androstenedione or dehydroepiandrosterone within the previous 4 weeks.
17. Has known malabsorption syndrome and/or current treatment with oral lipase inhibitors (eg, orlistat [Xenical®]) and/or bile acid-binding resins (eg, cholestyramine [Questran®], colestipol [Colestid®]) or treatments that promote gastric emptying (eg, metoclopramide [Reglan®]).
18. Inability to observe all rules and smoking restrictions in place at the clinical facility during confinement.
19. Has history of abuse of alcohol or any drug substance within the previous 2 years.
20. Poor compliance or unlikely to keep clinic appointments and remain for entire confinement period.
21. Has received any drug as part of another research study within 30 days of initial dose administration in this study.
22. Donated blood (≥ 500 mL) within the 12-week period before the initial study dose.
23. Current use of the following groups of drugs that effect T levels, T metabolism or levels of T metabolites, namely antiandrogens, 5-alpha-reductase inhibitors (eg, dutasteride, finasteride), estrogens, long-acting opioid analgesics (eg, methadone hydrochloride, buprenorphine hydrochloride) or human growth hormone (HGH).
24. Unwilling or unable to follow the dietary requirements for this study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01-21 (Actual); Study Completion 2017-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Swerdloff, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (2):
- United States (2):
  - Harbor-UCLA Medical Center, Torrance, California
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Testosterone Undecanoate 237 mg BID: Subjects complete Sequence A-E. Amount of Fat Varies by Sequence. Oral Testosterone Undecanoate 237 mg administered twice daily immediately prior to breakfast and immediately prior to dinner.
Period: Sequence A: Fasting
Arm/Group | Oral Testosterone Undecanoate 237 mg BID
Started | 18
Completed | 18
Not Completed | 0
Period: Sequence B: 15 g Fat Breakfast
Arm/Group | Oral Testosterone Undecanoate 237 mg BID
Started | 18
Completed | 18
Not Completed | 0
Period: Sequence C: 30 g Fat Breakfast
Arm/Group | Oral Testosterone Undecanoate 237 mg BID
Started | 18
Completed | 18
Not Completed | 0
Period: Sequence D: 45 g Fat Breakfast
Arm/Group | Oral Testosterone Undecanoate 237 mg BID
Started | 18
Completed | 18
Not Completed | 0
Period: Sequence E: FDA High Fat Breakfast
Arm/Group | Oral Testosterone Undecanoate 237 mg BID
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Oral Testosterone Undecanoate: Oral Testosterone Undecanoate 237 mg administered twice daily immediately prior to breakfast and immediately prior to dinner.
  Oral Testosterone Undecanoate
Arm/Group | Oral Testosterone Undecanoate
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Serum testosterone at screening (ng/dL) [Mean (Standard Deviation); unit: ng/dL] | 109.7 (85.98)

OUTCOME MEASURES:

1. Primary Outcome: Cmax-am for Oral TU Across Breakfast With Varying Fat Content
Description: Peak Concentration after morning dose (Cmax) for oral testosterone undecanoate taken after a fasting breakfast of varying fat content.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | Breakfast A - Fasting | Breakfast B - 15 g Fat | Breakfast C - 30 g Fat | Breakfast D - 45 g Fat | Breakfast E - High Fat
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
ng/dL | 250.7 (48.6) | 334.7 (57.7) | 529.7 (33.9) | 506.0 (37.8) | 463.4 (62.7)

2. Primary Outcome: Time of Peak Concentration (Tmax-am)
Description: The time of peak concentration (Tmax-am) will be assessed within each relevant dosing interval.
Time Frame: 12 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Breakfast A - Fasting | Breakfast B - 15 g Fat | Breakfast C - 30 g Fat | Breakfast D - 45 g Fat | Breakfast E - High Fat
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
hours | 4.000 [0.00 to 4.17] | 2.000 [0.00 to 11.92] | 2.000 [1.83 to 6.00] | 2.000 [1.92 to 11.92] | 2.000 [0.00 to 6.00]

3. Primary Outcome: Area Under the Curve (AUC-am)
Description: The 12 hours following morning dose area under the curve (AUC) will assessed for each sequence of breakfasts with varying fat content.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/dL
Arm/Group | Breakfast A - Fasting | Breakfast B - 15 g Fat | Breakfast C - 30 g Fat | Breakfast D - 45 g Fat | Breakfast E - High Fat
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
ng*hr/dL | 1905 (45.2) | 2428 (51.3) | 3279 (33.6) | 3395 (34.7) | 3187 (52.8)

4. Primary Outcome: Time Weighted Average Total Testosterone Concentration (Cavg-am)
Description: The time weighted average of total testosterone concentration will be assessed for each dosing interval.
Time Frame: 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | Breakfast A - Fasting | Breakfast B - 15 g Fat | Breakfast C - 30 g Fat | Breakfast D - 45 g Fat | Breakfast E - High Fat
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
ng/dL | 160.0 (45.4) | 203.7 (51.3) | 275.1 (33.6) | 285.1 (34.7) | 267.3 (52.6)

ADVERSE EVENTS:
Time Frame: Three months
Groups:
- Oral Testosterone Undecanoate 237 mg BID: Subjects will self-administer 237 mg oral TU BID for a 14 day Run-in Phase, followed by 5 consecutive days of twice daily dosing in a phase 1 clinic for serial PK sampling.
Arm/Group | Oral Testosterone Undecanoate 237 mg BID
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Testosterone Undecanoate 237 mg BID (N=18)
iron deficiancy anemia (Blood and lymphatic system disorders) | 1 (1)
abdominal pain upper (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
chest pain (General disorders) | 1 (1)
pyrexia (General disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 1 (1)
prostatic specific antigen increased (Investigations) | 1 (1)
white blood cell count increased (Investigations) | 1 (1)
headache (Nervous system disorders) | 1 (1)
dysuria (Renal and urinary disorders) | 1 (1)
pollakiuria (Renal and urinary disorders) | 1 (1)
prostatitis (Reproductive system and breast disorders) | 1 (1)
prostatomegaly (Reproductive system and breast disorders) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT02921386/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT02921386/SAP_001.pdf